CLINICAL TRIAL: NCT02299037
Title: Predicting the Risk of Post-operative Delirium: Use of Neuropsychology, Serum and CSF Biomarkers and Genetics to Predict Risk of Post-operative Delirium
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Belfast Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Dr Emma Cunningham, Clinical Lecturer Geriatric Medicine, Belfast Health and Social Care Trust
Other Study IDs: 09069PP-OPMS
Record Dates: First submitted 2014-10-31; First posted 2014-11-24 (Estimated); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum cerebrospinal fluid DNA extracted from blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to determine if pre-operative neuropsychological characteristics, apolipoprotein E4 status and/or cerebrospinal fluid (CSF) and serum biomarkers can predict those most at risk of post-operative delirium. Patients over the age of 65 years undergoing elective primary hip or knee arthroplasty in Musgrave Park Hospital are invited to take part. Participants undergo a pre-operative neuropsychological assessment which is repeated 6-12 weeks post-operatively at the time of surgical review appointment. At the time of surgery advantage is taken of the necessary venous cannulation and spinal anaesthetic to gain venous blood and CSF samples respectively. Venous blood is also sampled post-operatively. Patients are assessed daily for delirium, using the Confusion Assessment Method, until discharge. The association between delirium and subsequent cognitive decline is now well established in the literature. It is not yet clear whether this is solely because delirium following elective surgery indicates a previously unrecognised neurodegenerative process or whether the delirium itself exerts an additional pathophysiological insult. In order to investigate this, a follow-up study of these participants, approximately 8 years later is currently being conducted. Neuropsychological assessment and venous blood sampling will be repeated with consenting participants. Furthermore, the significance of subtle symptoms, not sufficient to fulfil the criteria for delirium and known as subsyndromal delirium, in relation to cognitive function years later will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* living at home
* undergoing primary, elective hip or knee arthroplasty
* spinal anaesthetic with intrathecal diamorphine anticipated

Exclusion Criteria:

* neurological, hearing or visual disability affecting ability to participate in study
* known neurodegenerative condition eg dementia, Parkinson's disease, multiple sclerosis

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients 65 years of age or more undergoing primary, elective hip and knee arthroplasty in a single surgical unit.
Sampling Method: Non-Probability Sample
Enrollment: 316 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-02 (Actual); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of inpatient post-operative delirium as measured using the confusion assessment method (CAM) | Day 1 post-operatively
Incidence of inpatient post-operative delirium as measured using the confusion assessment method (CAM) | Day 2 post-operatively
Incidence of inpatient post-operative delirium as measured using the confusion assessment method (CAM) | Day 3 post-operatively
Performance on the Mini-Mental Status Examination (MMSE; Folstein MF, Folstein SE et al. 1975). | 8 year follow-up
  A 30 point scale pre-operatively and at follow-up 7-8 years later.
Performance on the Executive Clock Drawing Task (CLOX 1 & 2; Royall, Cordes et al. 1998). | 8 year follow-up
  A 24 point scale pre-operatively and at follow-up 7-8 years later.
Performance on the Controlled Oral Word Association Test (COWAT; Benton, A.L. Hamsher, K. Sivan, A.B. 1983). | 8 year follow-up
  A test which measures both phonemic and semantic fluency. One point is awarded for each word generated (within the task parameters) within one minute. A total of five categories are assessed. Performance pre-operatively and at follow-up 7-8 years later will be compared.
Performance on the Stroop Colour and Word Test (Golden 1978). | 8 year follow-up
  This test features 100 items, the score reflects how many words were correctly identified in 45 seconds. A total of five categories are assessed. Performance pre-operatively and at follow-up 7-8 years later will be compared.
Colour Trails 1&2 (D'Elia, Satz et al. 1996). | 8 year follow-up
  Performance is measured in the time taken (seconds) taken to successfully complete this test. Performance pre-operatively and at follow-up 7-8 years later will be compared.
New York Paragraph Recall Test (Kluger, Ferris et al. 1999). | 8 year follow-up
  This test is scored based on the number of correctly recalled sections of the story. There are two recall conditions - immediate recall, assessed immediately following the reading of the paragraph and delayed recall, performance assessed five minutes following conclusion of the story. Each condition can earn a maximum of 21 points. Performance pre-operatively and at follow-up 7-8 years later will be compared.
Weighted Composite Summary Cognitive Measure at 7-8 year Follow-up | 8 year follow-up
  This weighted composite summary cognitive measure will be calculated based on the work of Inouye et al (Inouye, Marcantonio et al. 2016). This will be calculated (using outcome measures 4-9 above), for two time points 1) using preoperative scores and 2) using follow-up study visit scores. With the follow-up study visit scores being our primary outcome measure. The cognitive tests used in this study are similar to those utilised by the General Cognitive Performance score (Jones, Rudolph et al. 2010) and in deriving these scores we intend to use locally available normative data from representative samples, namely the Irish longitudinal studies (The Northern Ireland Cohort for the Longitudinal Study of Ageing (NICOLA) and The Irish Longitudinal Study on Ageing (TILDA)).

SECONDARY OUTCOMES:
Performance on the Mini-Mental Status Examination (MMSE; Folstein MF, Folstein SE et al. 1975). | 6-12 weeks post-surgery
  Performance on this 30 point scale pre-operatively and at follow-up 6-12 weeks later will be compared.
Performance on the Executive Clock Drawing Task (CLOX 1 & 2; Royall, Cordes et al. 1998). | 6-12 weeks post-surgery
  Performance on this 24 point scale pre-operatively and at follow-up 6-12 weeks later will be compared.
Performance on the Controlled Oral Word Association Test (COWAT; Benton, A.L. Hamsher, K. Sivan, A.B. 1983). | 6-12 weeks post-surgery
  A test which measures both phonemic and semantic fluency. One point is awarded for each word generated (within the task parameters) within one minute. A total of five categories are assessed. Performance pre-operatively and at follow-up 6-12 weeks later will be compared.
Performance on the Stroop Colour and Word Test (Golden 1978). | 6-12 weeks post-surgery
  This test features 100 items, the score reflects how many words were correctly identified in 45 seconds. A total of five categories are assessed. Performance pre-operatively and at follow-up 6-12 weeks later will be compared.
Colour Trails 1&2 (D'Elia, Satz et al. 1996). | 6-12 weeks post-surgery
  Performance is measured in the time taken (seconds) taken to successfully complete this test. Performance pre-operatively and at follow-up 6-12 weeks later will be compared.
New York Paragraph Recall Test (Kluger, Ferris et al. 1999). | 6-12 weeks post-surgery
  This test is scored based on the number of correctly recalled sections of the story. There are two recall conditions - immediate recall, assessed immediately following the reading of the paragraph and delayed recall, performance assessed five minutes following conclusion of the story. Each condition can earn a maximum of 21 points. Performance pre-operatively and at follow-up 6-12 weeks later will be compared.
Weighted Composite Summary Cognitive Measure at 6-12 Week Follow-Up | 6-12 weeks post-surgery
  This weighted composite summary cognitive measure will be calculated based on the work of Inouye et al (Inouye, Marcantonio et al. 2016). This will be calculated (using outcome measures 11-16 above), for two time points 1) using preoperative scores and 2) using follow-up study visit scores at 6-12 weeks post-operatively. With the follow-up study visit scores being our primary outcome measure. The cognitive tests used in this study are similar to those utilised by the General Cognitive Performance score (Jones, Rudolph et al. 2010) and in deriving these scores we intend to use locally available normative data from representative samples, namely the Irish longitudinal studies (The Northern Ireland Cohort for the Longitudinal Study of Ageing (NICOLA) and The Irish Longitudinal Study on Ageing (TILDA)).
Incidence of mild cognitive impairment and dementia at the time of follow-up study visit | 8 year follow-up
  Diagnosed using appropriate criteria (Albert, DeKosky et al., 2011, McKhann, Knopman et al., 2011).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Public Health, Queen's University Belfast, Belfast, United Kingdom